CLINICAL TRIAL: NCT06344429
Title: Exploring the Effects of Treatment With Stellest Lenses and Low-concentration Atropine for Myopia Control Among Children.
Brief Title: Stellest Lenses and Low-concentration Atropine Myopia Control Among Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Essilor-Polylite Taiwan Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STL_CT_0001
Record Dates: First submitted 2024-03-20; First posted 2024-04-03 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stellest lenses spectacle (Experimental): 34 children wear Stellest lenses for all day.
  Interventions: Device: Stellest Lenses
- Stellest lenses+0.05% atropine (Experimental): 33 children wear Stellest lenses for all day, and 0.05% atropine eye drops is dropped once nightly in both eyes.
  Interventions: Combination Product: Stellest Lenses+0.05% atropine
- Single vision lenses+0.05% atropine (Placebo Comparator): 33 children wear Single lenses for all day, and 0.05% atropine eye drops is dropped once nightly in both eyes.
  Interventions: Drug: Single vision Lenses+0.05% atropine

INTERVENTIONS:
Device: Stellest Lenses — All subjects are recruited and randomized to 3 treatment groups at the baseline visit.
  A Group：Stellest Lenses spectacle (ST)
  Arms: Stellest lenses spectacle
Combination Product: Stellest Lenses+0.05% atropine — All subjects are recruited and randomized to 3 treatment groups at the baseline visit.
  B Group：Combined Treatment
  Arms: Stellest lenses+0.05% atropine
Drug: Single vision Lenses+0.05% atropine — All subjects are recruited and randomized to 3 treatment groups at the baseline visit.
  C Group：0.05% Atropine with single vision
  Arms: Single vision lenses+0.05% atropine

SUMMARY:
The prevalence of myopia is increasing globally, especially in Asian countries. 70-80% of the young population suffers from myopia, and almost 20% have high myopia. High myopia can easily lead to blinding diseases, including retinal detachment, macular degeneration, and glaucoma. In Taiwan, according to a survey by the National Health Administration, the proportion of myopia among Grade 1 students has exceeded 81%.

There are many ways to control myopia progression. High concentrations of atropine have been reported highly effective in the control of the myopia progression. However the accompanied side effects such as photophobia and near blurred vision. Recent research shows that low-concentration atropine can achieve similar control effect and more acceptable with much minimal side effect compared to high concentration of atropine.

Multiple animal experiments have confirmed that giving retinal myopia defocus signals can effectively decrease the growth of the eye, thereby inhibiting the progression of myopia. Therefore, regarding lens design, myopic defocus does play an important role in myopia control, including orthokeratology lenses, multifocal soft contact lenses, and peripheral defocus lenses.

Stellest, a myopia control lens based on the myopia defocus theory, is equipped with highly aspheric lenslet technology. In a recent study, compared with single vision lenses, Stellest significantly slowed down the myopia progression reaching 67% and retard axial elongation reaching 64% The purpose of this study is to explore the effectiveness of Stellest Lenses in controlling myopia in Taiwanese children and whether Stellest Lenses combined with low-concentration atropine eye drops can increase the effect of myopia control.

DETAILED DESCRIPTION:
The prevalence of myopia has been increasing in the world, especially in East Asia. The prevalence of myopia and high myopia is estimated up to 50% and 10% of the global population, respectively in 2050. The social economic burden of this myopia epidemic will increase substantially, because of the risk of myopia-related complications, such as early onset of cataract, glaucoma, myopic macular degeneration and retinal detachment. The use of myopia control interventions in school myopia can help reduce severity of myopia in the further life of this population with potential reduce of the risk of these pathologies.

There are several ways to control school myopia progression. High concentrations of atropine have been reported highly effective in the control of the myopia progression. However the accompanied side effects such as photophobia and near blurred vision. Recent research shows that low-concentration atropine can achieve similar control effect and more acceptable with much minimal side effect compared to high concentration of atropine.

Research in animal models has shown that imposed myopic optical defocus in peripheral retina, the focal plane in front of the retina, has an inhibitory effect on eye growth to stop myopia progression. Recently, it has been reported that spectacle lenses with aspherical lenslets with myopic defocus (Stellest™ lenses) effectively slow myopia progression reaching 67% and retard axial elongation reaching 64% compared with single vision lenes in 1 year study.

The purpose of this study is to compare the effect of the Stellest lenses, 0.05% atropine and combined treatment for the myopia control in Taiwanese children.

Method： This study will be conducted 2 years at the Kaohsiung Chang Gung Memorial Hospital, Taiwan. Children aged 6 to 12 years old with myopic refraction of at least -0.75 D in both eyes, astigmatism of less than -2.5 D, were enrolled in this open label, randomized study. Excluded were those with ocular diseases (e.g., cataract, congenital retinal diseases, amblyopia, and strabismus), previous use of atropine, or orthokeratology lens orother optical methods for myopia control within 6 months, allergy to atropine, or systemic diseases (e.g., endocrine, cardiac, and respiratory diseases). Written informed consent will be obtained from parents or guardians and the participants. The study will be sent to the Ethics Committee of the Chang Gung Memorial Hospital and will be registered with the ClinicalTrials.gov Registry, the Kaohsiung Chang Gung Memorial Hospital (registration no:). All procedures are conducted according to the tenets of the Declaration of Helsinki.

100 Participants in this study were randomized to receive Stellest lenses spectacle (ST) (N=34), 0.05% atropine with single vision lenses (ASV) (N=33) and combined treatment (STA) (N=33). 0.05% atropine eye drops is dropped once nightly in both eyes in ASV and STA group. The gender and age are balanced across the 3 treatment arms. The trial medications were prepackaged identically with the number of study subjects and the expiration date. Expiry duration for the batch of eye drops was 2 years.

All subjects are recruited and randomized to 3 treatment groups at the baseline visit. Boys and girls are recruited to have a balance in gender. All subjects are then followed up on the same schedule with the same examination protocol: at 2 weeks (monitor visit), 6 months, and 12 months from the baseline visit. The purpose of the monitor visit at 2 weeks was to determine the hyperopic shift, if any, that has been reported in a higher concentration of atropine in the previous studies.

At each visit, distant best-corrected visual acuity (BCVA) in was assessed by an optic technician using the Landolt C chart and Optical Coherence Tomography (OCT) by well-trained an study team staff. Near visual acuity was assessed using best-corrected distance spectacle correction with a reduced logMAR reading chart placed at 40 cm under well-lit conditions. The near point of accommodation was measured using a Royal Air Force (RAF) near point rule (Harlow, Essex, UK) with best-corrected distance spectacle correction.

Participants were instructed to move the target inward until the N5 print became slightly blurred and then outward until it just became clear. Accommodation amplitude was calculated as the inverse of the near point of accommodation.

Mesopic pupil size and photopic pupil size were measured. Cycloplegic autorefraction was performed using an autorefractor after the tropicamide regimen, which consisted of at least 3 cycles of eye drops. At the first cycle, 2 separate eye drops, tropicamide 1%, were administered to both eyes at 5 minutes apart. A 2nd and 3rd cycle of the same cycloplegic drops would be administered 10 minutes after the previous cycle. If the pupil size was less than 6.0 mm, further cycles of cycloplegic eye drops would be administered if necessary to ensure the pupils are well dilated. Five readings, all of which had to be less than 0.25 D apart, were obtained and averaged. Spherical equivalent (SE) was calculated as spherical power plus half of the cylinder power. Ocular AL was measured by on noncontact partial coherence interferometry and optic coherencetomography. Five readings, with a maximum-minimum deviation of 0.05 mm or less, were taken and averaged. A diary on the trial medication was kept for each subject. Compliance level of each subject was classified according to the mean number of using atropine per week as reported by participants over the 12 months. Subjects with 75% compliance rate (i.e., a mean of 5.25 days/week) were considered to have good compliance. Subjects were also offered sunwear orsunglasses or (which darken on exposure to ultraviolet or sunlight) if they experienced glare or if their parents were worried of excessive light exposure, or progressive glasses (reading add) if they experienced difficulty with near vision. All subjects were prescribed with best-corrected spectacles.

At the baseline, validated questionnaires on outdoor time and near work were administered to parents. In addition, children wear outdoor time smartwatch for 1 week to evaluation the outdoor time every day in the baseline, 6-month F/U and 12-month F/U. Outdoor activities includes time spent on sports and leisure, whereas near works included time on homework, cell phone, computer, video games, and watching TV. Parental refraction is documented by noncycloplegic autorefraction measurement, for both parents of each child at baseline. At the 12-month follow-up visit, the Chinese version of the 25-Item National Eye Institute Visual Function Questionnaire was administered to all subjects to determine the impact of different treatment groups on the vision-related quality of life.

A total of 11 subscales are addressed: general health, general vision, ocular pain, near vision, distance vision, social function, mental health, role limitations, dependency, color vision, and peripheral vision. Driving is excluded.

The primary outcome was myopia progression in terms of SE change over 1 year. Myopia progression in each eye was further categorized as mild (<0.5 D), moderate (0.5-0.99 D), or severe (≥1.0 D). The secondary outcomes included AL change at 1 year. Side effect parameters included changes in accommodation amplitude, mesopic and photopic pupil sizes, and distant BCVA and near visual acuity. All ophthalmic parameters, including SE, AL, accommodation, pupil size, and visual acuity, were monitored from baseline.

During each visit, subjects and parents were given an open-ended opportunity to report any medical illness or adverse events. They were also specifically asked about symptoms related to allergy, blurred near vision, glare, or visual loss, and if subjects had been ill or hospitalized since the previous visit. Adverse events (AEs) will be followed, recorded, and reported in the CRF throughout the entire study and only relevant to spectacle or atropine used signs and symptoms. The investigator will assess the severity (intensity) of each AE as mild, moderate or severe, and will also categorize each AE as to its potential relationship to IP (0.05% atropine or Stellest Lenses) using the categories of yes or no.

An Serious Adverse Events (SAE)，an SAE is any event that meets any of the following criteria: Results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/ birth defect, is important medical event. Investigator is obliged to respond and meet strict regulatory and IRB timelines associated with expedited reporting obligations for events of this nature. Relevant SAE reporting and follow up information should be notice sponsor immediately and file it along.

Confidentiality and Data Management All information generated in this study is considered highly confidential and must not be disclosed to any person or entity directly involved with the study unless prior written consent is gained from the sponsor. However, authorized regulatory officials, IRB personnel, the sponsor, and its authorized representatives are allowed full access to the records.

All study subjects and legal representative must be informed that their personal study-related data will be used by the sponsor in accordance with local data protection law and the General Data Protection Regulation. The level of disclosure must also be explained to the subject and legal representative, who will be required to give consent for their data to be used as described in the ICF. The subject and legal representative must be informed that medical records may be examination by auditors or other authorized personnel appointed by the sponsor, by appropriated IRB members, and by inspectors from regulatory authorities.

Identification of subjects and CRFs shall be by unique subject identification numbers only. All personal identifiers according to applicable regulations (eg, number, phone number) must be redacted permanently by the site personnel and replaced with the subject's unique identification member in all records and data before transfer to the sponsor (or designee).

All personnel details will be treated as confidential by the investigator and staff.

Statistical Analysis： All data were analyzed based on the intention-to-treat principle. Change of parameters was defined by the difference between the baseline and the corresponding follow-up values. Chi-square test and Fisher exact test were used to test the group difference in categoric data. Analysis of variance was used to test the group difference of continuous data. SPSS software was used for data analyses. P value < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 6~12 year-old.
2. Equivalent diopter: -0.75~-4.00 D.
3. Astigmatism and anisometropia <2.50 D.
4. Best corrected visual acuity of one eye reaches 1.0.

Exclusion Criteria:

1. Strabismus, amblyopia, and abnormal binocular vision.
2. Other eye diseases.
3. Have a history of using myopia control products within six months.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2024-08-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Spherical equivalent refraction power | At 2 weeks (monitor visit), 6 months, and 12 months from the baseline visit
  Spherical equivalent (SE) was calculated as spherical power plus half of the cylinder power
Axial length | At 2 weeks (monitor visit), 6 months, and 12 months from the baseline visit
  Ocular AL was measured by on non contact partial coherence interferometry and optic coherence tomography.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan